CLINICAL TRIAL: NCT06986057
Title: Iparomlimab and Tuvonralimab (QL1706) Combined With Platinum-Based Chemotherapy for Neoadjuvant Treatment of Cervical Cancer: A Single-Arm Phase II Clinical Trial
Brief Title: Iparomlimab and Tuvonralimab Combined With Platinum-Based Chemotherapy for Neoadjuvant Treatment of Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Tumor Hospital (Other)
Responsible Party: Principal Investigator, Dapeng Li, Principal Investigator, Shandong Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-CC-IIT-003
Record Dates: First submitted 2025-04-16; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer; Neoadjuvant Therapy
Keywords: immunotherapy; PD-1 Inhibitor; CTLA-4 Inhibitor
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Evaluation of the Efficacy of Iparomlimab and Tuvonralimab in Combination with Platinum-Based Chemotherapy for Neoadjuvant Therapy of Cervical Cancer
  Interventions: Drug: Iparomlimab and tuvonralimab (QL1706) combined with platinum-based chemotherapy

INTERVENTIONS:
Drug: Iparomlimab and tuvonralimab (QL1706) combined with platinum-based chemotherapy — Iparomlimab and tuvonralimab (QL1706) combined with platinum-based chemotherapy

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of Iparomlimab and tuvonralimab (QL1706) in combination with platinum-based chemotherapy for cervical cancer neoadjuvant therapy. Additionally, the study aims to identify potential predictive biomarkers for therapeutic efficacy by analyzing tumor tissues and peripheral blood samples from participants receiving this combined treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of written Informed Consent Form (ICF).
* Age ≥18 years and ≤75 years at enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Histologically or cytologically confirmed cervical cancer (squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma) with clinical staging by FIGO 2018 criteria: IB3, IIA2, IIB, or IIIC (parametrial invasion without reaching the pelvic wall, no vaginal lower third involvement).
* No prior systemic or local antitumor therapy (including radiotherapy, chemotherapy, immunotherapy, biologics, or small-molecule targeted therapy) for cervical cancer prior to the first dose of study treatment.

Agreement to undergo radical hysterectomy with no surgical contraindications as judged by the investigator.

* At least one untreated measurable lesion according to RECIST v1.1.
* Consent to provide tumor tissue and peripheral blood samples during the screening period and study procedures for related research.
* Adequate organ function:

  a) Hematology (no blood components or growth factor support within 7 days before study treatment): i. Absolute neutrophil count (ANC) ≥1.5×10⁹/L (1,500/mm³); ii. Platelet count ≥100×10⁹/L (100,000/mm³); iii. Hemoglobin ≥90 g/L. b) Renal: i. Calculated creatinine clearance (CrCl) ≥50 mL/min (Cockcroft-Gault formula); ii. Urine protein <2+ or 24-hour urine protein <1.0 g. c) Hepatic: i. Total bilirubin (TBil) ≤1.5×ULN; ii. AST and ALT ≤2.5×ULN; iii. Albumin (ALB) ≥28 g/L. d) Coagulation: i. INR and APTT ≤1.5×ULN (stable anticoagulation therapy allowed if parameters remain within therapeutic range).

  e) Cardiac: i. Left ventricular ejection fraction (LVEF) ≥50%.
* Fertile women must have a negative urine or serum pregnancy test within 3 days before first dose. If urine test is inconclusive, serum testing is required. Contraception must be used from screening until 120 days post-treatment. Barrier methods or hormonal contraceptives (e.g., pills) are required.

  1. Fertile women: Not surgically sterilized (e.g., bilateral tubal ligation) or premenopausal (≥12 months amenorrhea with FSH in postmenopausal range).
  2. Effective contraception: Methods with <1% failure rate (e.g., hormonal contraceptives).
* Willingness and ability to comply with scheduled visits, protocols, labs, and study requirements.
* Expected survival ≥6 months.

Exclusion Criteria:

* Histopathological type other than cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma (e.g., small cell carcinoma, clear cell carcinoma, sarcoma).
* History of other malignancies within 3 years prior to enrollment, excluding localized malignancies cured by local therapy (e.g., basal cell carcinoma, squamous cell carcinoma of the skin, or ductal carcinoma in situ of the breast).
* Simultaneous enrollment in another clinical study, unless it is an observational, non-interventional study or within the follow-up period of an interventional study.
* Non-specific immunomodulatory therapy (e.g., interleukins, interferons, thymosin, tumor necrosis factor) within 2 weeks prior to first dose; herbal or proprietary Chinese medicine with antitumor indications within 1 week prior to first dose.
* Active autoimmune disease requiring systemic therapy (e.g., disease-modifying agents, corticosteroids, immunosuppressants) within the past 2 years. Replacement therapy (e.g., thyroid hormone, insulin, or physiological corticosteroids for adrenal/pituitary insufficiency) is not considered systemic therapy.
* History of non-infectious pneumonia requiring systemic corticosteroids or current interstitial lung disease.
* Significant bleeding diathesis or coagulation dysfunction.
* Uncontrolled comorbidities, including but not limited to decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease/gastritis, or psychiatric/social conditions impairing compliance or informed consent.
* History of myocarditis, cardiomyopathy, or malignant arrhythmias. Within 12 months prior to first dose: unstable angina, congestive heart failure, or vascular disease requiring hospitalization (e.g., surgical repair of aortic aneurysm/peripheral venous thrombosis). Within 6 months prior: esophageal-gastric varices, unhealed wounds, gastrointestinal perforation, fistula, obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding. Arterial thromboembolism, NCI CTCAE 5.0 grade ≥3 venous thromboembolism, transient ischemic attack, stroke, hypertensive crisis, or hypertensive encephalopathy. Within 1 month prior: acute exacerbation of COPD. Current hypertension uncontrolled with oral antihypertensives (SBP ≥160 mmHg or DBP ≥100 mmHg).
* Active or history of definite inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea).
* Severe infection within 4 weeks prior to first dose (including hospitalization, sepsis, or severe pneumonia). Active infection requiring systemic antimicrobial therapy within 10 days prior (excluding HBV/HCV antiviral therapy).
* Major surgery or severe trauma within 30 days prior to first dose; minor local procedures (excluding peripherally inserted central catheter placement) within 3 days prior.

History of immunodeficiency, HIV seropositivity, or current long-term systemic corticosteroid/immunosuppressant use.

* Active pulmonary tuberculosis (TB) or suspected TB requiring clinical exclusion (e.g., sputum AFB, chest X-ray).
* Active syphilis infection.
* History of allogeneic organ or hematopoietic stem cell transplantation.
* Untreated active HBV (HBsAg+ with HBV-DNA >1000 copies/mL [200 IU/mL] or above limit of detection). HBV patients must receive antiviral therapy during study. Active HCV (HCV Ab+ with HCV-RNA above limit of detection).
* Live vaccine administration within 30 days prior to first dose or planned during study.
* Known hypersensitivity to any study drug component or severe allergic reaction to other monoclonal antibodies.
* History of psychiatric disorders, substance abuse, alcoholism, or drug addiction.
* Pregnancy or lactation.
* Any disease, treatment, or laboratory abnormality that may confound study results, hinder compliance, or compromise participant safety.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CR/PR rate (%) in subjects with ≥1 response event | 4 months after the patient was enrolled in the study
  The ORR assessment will include data obtained before surgery or until disease progression (whichever occurs first), or until the last evaluable assessment data before surgery if no disease progression has occurred.

SECONDARY OUTCOMES:
pCR rate (%) post neoadjuvant therapy | 6 months after the patient was enrolled in the study
  The proportion of patients with no residual tumor cells in the tumor tissue specimens obtained through surgical resection after neoadjuvant therapy.
Time to first event post-neoadjuvant therapy | 2 years after the patient was enrolled in the study
  The time from the start of neoadjuvant therapy to the occurrence of any of the following events for the patient: disease progression, local or distant recurrence diagnosed by imaging or biopsy, death due to any cause, etc.
Patients whose residual active tumor cells are ≤ 10% after neoadjuvant therapy | 6 months after the patient was enrolled in the study
  MPR（Major Pathological Response） rate = (Number of subjects achieving MPR / Total number of subjects) × 100%.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2 years after the patient was enrolled in the study
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Surgical Delay Rate (%) | 6 months after the patient was enrolled in the study
  rate = delayed cases / total cases × 100%

IPD SHARING:
Plan to Share IPD: Undecided